CLINICAL TRIAL: NCT06015997
Title: The Prevalence of ATTR Cardiac Amyloidosis in Elderly Middle Eastern Patients Undergoing Transarterial Aortic Valve Replacement
Brief Title: Prevalence of ATTR Cardiac Amyloidosis in Patients Undergoing TAVR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: ANAC.JO.2023.ATTR.TAVR.ME
Record Dates: First submitted 2023-08-23; First posted 2023-08-29 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: ATTR Amyloidosis Wild Type; Severe Aortic Stenosis; Aortic Valve Stenosis; Middle East Studies
Keywords: ATTR cardiac amyloidosis; Severe aortic stenosis; Transarterial aortic valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ATTR-cardiac amyloidosis (CA) is present in 4% to 16% of elderly patients with severe calcific aortic stenosis (AS). The reasons for this association are not fully known. It is hypothesized that an amyloidotic infiltration of the aortic valve acts as a trigger for the development of endothelial damage and subsequent calcification. Elderly patients undergoing TAVI will be evaluated for the presence of ATTR-CA in Jordan.

DETAILED DESCRIPTION:
ATTR-cardiac amyloidosis (CA) is present in 4% to 16% of elderly patients with severe calcific aortic stenosis (AS). The reasons for this association are not fully known. Two hypotheses may explain this association

1. Amyloidotic infiltration of the aortic valve acts as a trigger for the development of endothelial damage and subsequent calcification.
2. The increased myocardial strain induced by AS may locally favor the process of amyloidogenesis and tissue infiltration.

Transarterial AV replacement (TAVI) is the treatment of choice for elderly patients with severe calcific AS. Studies have shown a prevalence of about 10% of ATTR cardiac amyloidosis in patients undergoing TAVI. The diagnosis is based on a positive nuclear scan (PYP, DPD or HMDP) and ruling out AL amyloidosis in patients with positive scans. While studies have shown no impact of ATTR on prognosis in TAVI patients, there is evidence of poorer quality of life, increased in-hospital acute ischemic stroke, increased cardiac and heart failure hospitalizations, increased conduction abnormalities, compared to patients without ATTR undergoing TAVI.

The prevalence of ATTR in TAVI patients in Jordan and Middle Eastern populations has not been previously evaluated. The purpose of this study is to evaluate the prevalence of ATTR cardiac amyloidosis in elderly Middle Eastern patients undergoing TAVI and to document the clinical characteristics, procedural outcomes and 1 year follow up of such patients compared to patients without ATTR.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Severe aortic stenosis
* Patient underwent TAVR procedure
* Positive pyruvate PO4 scan

Exclusion Criteria:

* Diagnosis of AL amyloidosis base on free light chain assay, serum and urine immune electrophoresis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Consecutive elderly patients, 65 years of age or older, with a diagnosis of severe aortic stenosis who undergo TAVR will be evaluated for the possible diagnosis of an underlying ATTR cardiac amyloidosis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence of ATTR CA in TAVR patients | On admission ( from time of admission to time of discharge from the hospital) and within 10 days.
  Consecutive elderly (≥65 years) patients who are undergoing TAVI will be included.
  Patients will be invited to undergo a pyruvate PO4 (PYP) scan. Patients with positive scans will undergo further testing to rule out AL amyloidosis (Free light chain assay, SIFEP, UIFEP). Data collection will include all pertinent clinical characteristics, peri- procedural details.
Cardiovascular event at One year follow up | One year after enrollment: up to 30 days after the passage of 365 days after the TAVR procedure
  Events at one year defined as the occurrence of all-cause death, and hospital admission for heart failure or aortic valve reintervention.